CLINICAL TRIAL: NCT06188806
Title: Investigation of the Effect of Proximal and Distal Adductor Canal Block on Pain Control and Functional Mobility in Total Knee Prosthesis Surgery Performed Under Spinal Anesthesia
Brief Title: Investigation of the Effect of Proximal and Distal Adductor Canal Block in Knee Replacement Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, head of Anesthesia and reanimation, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URH-AR-ZT-06
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: adduktor canal block,knee artroplasti,postoperative pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: three groups Group 1: proximal ACB (n:26) Group 2: distal ACB(n:26) Group 3: Control group (n:26)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PROXİMAL ADDUKTOR CANAL BLOCK GROUP (Active Comparator): Patients are placed in the supine position and a high-frequency linear probe is inserted for a cross-sectional image of the groin and thigh. The femoral nerve is identified in the short axis near the inguinal crease and the ultrasound transducer is placed caudally beyond the femoral triangle. The location of the proximal block is determined where the superficial femoral artery passes under the medial border of the sartorius muscle (usually 8-12 cm distal to the inguinal crease). Using the in-plane technique, a 100 mm peripheral nerve block needle is advanced until the tip of the needle passes the sartorius muscle and enters the adductor canal from the lateral side of the superficial femoral artery, and 20 mL 0.375% Bupivacaine is administered. To verify block success, sensory function is assessed by pinprick testing along the saphenous nerve distribution by comparing the pinprick sensation to the unaffected limb.
  Interventions: Other: ADDUKTOR CANAL BLOCK
- DİSTAL ADDUKTOR CANAL BLOCK GROUP (Active Comparator): Patients are placed in the supine position, the mid-thigh point is determined as half the distance between the groin crease and the top of the patella. After the mid-thigh mark is marked with a sterile marking pen, the ultrasound transducer is positioned for a transverse view of the adductor canal into the mid-thigh. Under USG imaging, the femoral artery and saphenous nerve are identified. The distal position is determined where the USG probe moves away from the sartorius muscle of the femoral artery and proceeds deep into the adductor hiatus, and a 100 mm block needle passes the sartorius muscle with an in plane technique and 20 mL 0.375% Bupivacaine is administered to the lateral side of the femoral artery and saphenous nerve.
  Interventions: Other: ADDUKTOR CANAL BLOCK
- CONTROL GROUP (Sham Comparator): No nerve block procedure is applied to patients.
  Interventions: Other: CONTROL GROUP

INTERVENTIONS:
Other: ADDUKTOR CANAL BLOCK — All patients who will undergo adductor canal block are sedated with midazolam 0.03 mg/kg in the preoperative preparation room, after standard monitoring. After 2-3 ml skin infiltration with 2% lidocaine under sterile conditions, a block is applied under USG guidance.To verify block success, sensory function is assessed by pinprick testing along the saphenous nerve distribution by comparing the pinprick sensation to the unaffected limb.All patients are monitored in the operating room and in a sitting position, 10-20 mg (2-4 ml) of heavy marcaine (0.5% bupivacaine hydrochloride and dextrose monohydrate) is applied to the subarachnoid space by entering the L3-4 or L4-5 space with a 25-gauge Whitrace needle.For postoperative multimodal analgesia, which is routinely applied to all patients, intravenous PCA (patient controlled analgesia )tramadol and paracetamol 10 mg / kg iv (8 hours apart) will be given.
  Arms: DİSTAL ADDUKTOR CANAL BLOCK GROUP; PROXİMAL ADDUKTOR CANAL BLOCK GROUP
Other: CONTROL GROUP — No nerve block procedure is applied to patients.All patients are monitored in the operating room and in a sitting position, 10-20 mg (2-4 ml) of heavy marcaine (0.5% bupivacaine hydrochloride and dextrose monohydrate) is applied to the subarachnoid space by entering the L3-4 or L4-5 space with a 25-gauge Whitrace needle.For postoperative multimodal analgesia, which is routinely applied to all patients, intravenous PCA (patient controlled analgesia) tramadol 50 mg at 10 mg / hour basal rate after loading (20 mg bolus dose + 30 minutes lock time) and paracetamol 10 mg / kg iv (8 hours apart) will be given.
  Arms: CONTROL GROUP

SUMMARY:
to investigate the effect of adductor canal block applied with two different approaches in the treatment of pain after TKA surgery on pain control and functional mobility.

DETAILED DESCRIPTION:
This prospective randomized trial is randomly divided into 3 groups using the method. Total knee arthroplasty is performed by the same surgical team.

is applied. The patients were divided into proximal ACB applied, distal ACB applied and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Medications for unilateral TKA surgery

  * Patients aged 18-85
  * ASA 1-3

Exclusion Criteria:

* Patients under 18 years of age and over 85 years of age
* Patients with ASA 4 and above
* Patients with cognitive impairment
* Patients with application site infection
* Patients allergic to local anesthesia
* Patients receiving anticoagulant therapy
* Patients with bleeding diathesis
* Patients with chronic opioid or substance use
* Patients with insulin-dependent diabetes mellitus
* patients with neuropathy

  * patients with hepatic or renal failure
* Patients who do not accept the procedure to be applied

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
VISUAL ANALOGUE SCALE(VAS) | POSTOPERATIVE 6, 12 AND 24 HOURS
  VAS pain score was evaluated as "no pain" (score=0) and "worst pain" (score=10) and was divided into 3 groups according to the World Health Organization's pain intensity scale: score <3 mild pain, 3-6 mild-moderate. degree pain and >6 moderate-severe pain.

SECONDARY OUTCOMES:
first mobilization time | within postoperative 24 hours
  The first postoperative mobilization hours of the patients will be recorded.
length of hospital stay | ONE WEEK
  The time between patients' admission and discharge will be recorded.
opioid use | within postoperative 24 hours
  Intravenous PCA will be applied to each patient and the total tramadol dose spent will be calculated.intravenous PCA (patient controlled analgesia) tramadol 50 mg at 10 mg / hour basal rate after loading (20 mg bolus dose + 30 minutes lock time)

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)